CLINICAL TRIAL: NCT01069042
Title: A Clinical Study on Anti-Hypertensive Agent (ACEi) and Heart Function Improvement
Brief Title: Anti-Hypertensive Agent (ACEi) and Heart Function Improvement in Association With Rho Kinase Activity Changes in Human
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Ping-Yen Liu, MD, PhD, Assistant Professor of Internal Medicine, National Cheng-Kung University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR-98-096
Record Dates: First submitted 2010-02-12; First posted 2010-02-17 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Heart Failure
Keywords: Rho kinase activity; Heart failure; ACE inhibitor; LVEF change; Rho kinase activity change
MeSH Terms: conditions — Heart Failure | interventions — Enalapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- preserved LVEF under ACEi treatment (Active Comparator): preserved LVEF under ACEi treatment
  Interventions: Drug: Enalapril
- Poor LVEF group (Experimental): Poor LVEF under ACEi treatment
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Enalapril — All subjects will initially receive 10mg of enalapril and be gradually titrated up to 20mg with blood pressure tolerance for 6 months.
  Other Names: Renitec

SUMMARY:
Hypothesis: Rho, one of the small GTPase proteins, and its downstream target molecule, Rho-kinase (ROCK), play important roles in mediating various cellular functions, including contractility, actin cytoskeleton organization, cell adhesion and motility, proliferation, cytokinesis and gene expressions, all of which are involved in the pathogenesis of cardiomyocyte contractility and other vascular disease. The investigators thus hypothesize that ROCK pathway plays an important role in the function and severity of heart failure (HF) and can be one of the possible pathway that currently applied cardiovascular medicine affecting their prognosis among HF treatment.

Previous study has shown that in patients with HF, intra-arterial infusion of fasudil causes preferential increase in forearm blood flow as compared with control subjects, suggesting an involvement of Rho/Rho-kinase pathway in the increased peripheral vascular HF failure remain to be examined. Besides, whether the rho kinase activity was enhanced or their response to current medication in HF patients remained unsolved.

Aim: ROCK activity and left ventricular function between HF or non-HF population survey and their response to ACEi Tx.

DETAILED DESCRIPTION:
Study design: We will enroll subjects from clinics of National Cheng Kung University Hospital.

Subjects will be then divided to two groups by their left ventricular ejection fraction (LVEF) ratio: preserved LVEF (EF>40%) and impaired LVEF (EF<40%). All subjects will initially receive 10mg of enalapril and be gradually titrated up to 20mg with blood pressure tolerance for 6 months. Before and after 6 months, echocardiography and blood sample will be assayed for biomarkers and rho kinase activity, respectively.

Outcomes and measurement: The outcomes will include the mean changes in the Rho-kinase activity in leukocytes before and after periods of treatment. Leukocyte Rho-kinase expression and activity will be measured in cells isolated from peripheral blood samples and frozen at -80 °C. The other outcomes are the correlation between the mean changes in Rho-kinase activity in leukocytes and cardiac function measured by 2D and M-mode echocardiography. In addition, we will calculate the association of ROCK activity and B-type natriuretic peptide (BNP), high sensitivity C-reactive protein (hsCRP) as well as its relation with clinical characteristics. The demographic, relevant clinical data and laboratory results will be all collected from patients and/or medical records.

Primary Outcomes and measurement: The primary outcomes are the mean changes in the Rho-kinase activity in leukocytes before and after periods of treatment. Leukocyte Rho-kinase expression and activity will be measured in cells isolated from peripheral blood samples and frozen at -80 °C. Western Blot assays will be performed to measure Rho-kinase activity .

Secondary Outcomes and measurement: The secondary outcomes are the correlation between the mean changes in Rho-kinase activity in leukocytes and cardiac function measured by echocardiography and tissue Doppler to measure systolic and diastolic function. In addition, the association of Rho kinase activity and BNP, hsCRP as well as its relation with clinical characteristics will be measured.

Besides, we will check the renal and liver function deterioration, changes in serum potassium levels, need for kidney replacement therapy and postural hypotension or dizziness or shock events to monitor the safety issues. Other parameters of adding medication will be recorded, including side effects like cough, angioedema, skin rash, intolerance to the medication.

ELIGIBILITY:
Inclusion Criteria:

* those subjects aged from 16 to 80 years
* diagnosed as systolic hypertension

Exclusion Criteria:

* renal insufficiency (serum creatinine ≥ 2.5 mg/dl)
* hyperkalemia (serum potassium ≥ 5mmol/L)
* with systemic inflammatory disease, including history of autoimmune disease, malignance; bilateral renal artery stenosis
* prior intolerance of an angiotensin receptor blockade (ARB) or ACE
* ACEi or ARB use within recent 1 month
* record of symptomatic hypotension

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-08 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
The primary outcomes are the mean changes in the Rho-kinase activity in leukocytes before and after periods of treatment. | 3 and 6 months

SECONDARY OUTCOMES:
The correlation between the mean changes in Rho-kinase activity in leukocytes and cardiac function measured by echocardiography. | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Hong Chen, MD, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan